CLINICAL TRIAL: NCT07090902
Title: Effect of Childbirth Preparation Education Using Progressive Relaxation Exercise on Birth Mode Preference, Labor Pain and Breastfeeding Comfort
Brief Title: The Effect of Progressive Relaxation Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Reyhan Aydin Doğan, Associate Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/1493; KBÜBAP-24-YL-010 (Other Grant/Funding Number: karabük üniversity)
Record Dates: First submitted 2025-06-20; First posted 2025-07-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Pregnancy; Labor Pain
Keywords: Progressive relaxation exercise; labor pain; delivery method; breastfeeding
MeSH Terms: conditions — Breast Feeding; Labor Pain

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized controlled trial with two arms: one intervention group receiving childbirth preparation training with progressive relaxation exercises, and one control group receiving standard prenatal care.
Masking Description: This is an open-label study. No masking is applied to participants, care providers, outcome assessors, or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Relaxation-Based Childbirth Preparation Program (Experimental): A structured education program including progressive muscle relaxation techniques delivered through face-to-face instruction, printed materials, and a guided CD. Participants are asked to follow daily exercises at home until birth.
  Interventions: Behavioral: Progressive Relaxation-Based Childbirth Preparation Program
- Control Group (No Intervention): Participants in this group will receive standard antenatal care provided by the hospital. No additional childbirth education or relaxation training will be offered.

INTERVENTIONS:
Behavioral: Progressive Relaxation-Based Childbirth Preparation Program — This intervention consists of a childbirth preparation program that integrates progressive muscle relaxation (PMR) exercises. Participants receive face-to-face education by trained health professionals, a printed booklet explaining both childbirth preparation and PMR techniques, and an audio CD with guided relaxation sessions produced by the Turkish Psychological Association. The participants are instructed to perform the relaxation exercises daily at home until delivery. The goal of this intervention is to reduce labour pain, support informed mode of delivery preference, and enhance breastfeeding comfort in the early postpartum period.
  Other Names: PMR-Enhanced Antenatal Program
  Arms: Progressive Relaxation-Based Childbirth Preparation Program

SUMMARY:
This clinical trial aims to evaluate the effect of a childbirth preparation program that includes progressive relaxation exercises on pregnant women's preferences for mode of delivery, their experience of labour pain, and breastfeeding comfort. Participants in the intervention group will receive a specially developed educational booklet and an audio CD with guided exercises, along with face-to-face training sessions. The control group will receive standard prenatal care. The study will help determine whether relaxation-based training can support women in coping with labour more comfortably and influence their choices and early postpartum experiences.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to evaluate the effectiveness of a childbirth preparation education program that incorporates progressive relaxation exercises. The intervention was developed to address the physical and psychological challenges pregnant women face, particularly in managing labour pain, making informed decisions about mode of delivery, and achieving comfort in early breastfeeding.

The study will be conducted in four stages. First, a childbirth preparation booklet including progressive relaxation techniques will be created based on current literature and expert guidance. Second, the content will be reviewed by a panel of experts to ensure content validity. Third, eligible pregnant women will receive in-person training sessions supported by the booklet and a relaxation exercise CD developed by the Turkish Psychological Association. Lastly, participants will be instructed to practice the exercises daily at home, and the effectiveness of the intervention will be evaluated using validated measurement tools.

The trial will be conducted in Samsun, Türkiye, and will include 40 pregnant women meeting specific inclusion criteria. Participants will be randomly assigned to either the intervention group or the control group. Outcomes will be measured using established scales such as the Visual Analogue Scale (VAS) for labour pain, LATCH for breastfeeding, and a postpartum comfort scale. The results of this study may contribute to the development of accessible, low-cost, and culturally appropriate childbirth education strategies in Türkiye and globally.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 18 and 49 years
* Currently pregnant
* Willing to participate in the study and provide informed consent
* Able to attend the planned training sessions regularly
* No complications during pregnancy, childbirth, or postpartum for themselves or their newborn

Exclusion Criteria:

* Not within the age range of 18-49
* Not currently pregnant
* Fails to complete study questionnaires or withdraws from the study
* Has communication difficulties or cognitive impairment
* Fails to attend training sessions regularly
* Has open wounds or allergic skin conditions
* Develops postpartum complications (e.g., bleeding, infection, fever)
* Has cardiac arrhythmia or uses a pacemaker
* Diagnosed with conditions such as epilepsy or pre-eclampsia
* Has kidney or liver disease
* Previously practiced progressive muscle relaxation techniques
* Is morbidly obese (BMI > 40)
* Uses chronic opioids, antidepressants, or psychoactive medications

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
During active labour (at 4-7 cm cervical dilation | within 5 hours after the start of labor
  Labour pain will be assessed using the Visual Analogue Scale (VAS), a 10-point self-reported pain scale. Higher scores indicate more intense pain.

SECONDARY OUTCOMES:
The type of birth and the type of birth they want during pregnancy. | 36-38 weeks of pregnancy and within 2 days after birth
  The preferred and actual mode of delivery (vaginal vs. caesarean section) will be recorded and compared between intervention and control groups.
Breastfeeding Comfort | Within 2 hours after delivery (Within 24 hours after delivery)
  Breastfeeding comfort will be evaluated using the Postnatal Comfort Scale
Pain Intensity Score | within 5 hours after the start of labor
  Pain intensity was measured using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Training and Research Hospital, Department of Obstetrics and Gynecology, Samsun, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sercekus P, Baskale H. Effects of antenatal education on fear of childbirth, maternal self-efficacy and parental attachment. Midwifery. 2016 Mar;34:166-172. doi: 10.1016/j.midw.2015.11.016. Epub 2015 Nov 27. PMID 26656473
- [Result] Liu K, Chen Y, Wu D, Lin R, Wang Z, Pan L. Effects of progressive muscle relaxation on anxiety and sleep quality in patients with COVID-19. Complement Ther Clin Pract. 2020 May;39:101132. doi: 10.1016/j.ctcp.2020.101132. Epub 2020 Mar 6. PMID 32379667